CLINICAL TRIAL: NCT05261711
Title: A Phase 1/2, Open-Label, Dose Escalating Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AB1 in Adult Patients with Sickle Cell Disease (SCD)
Brief Title: AB1 in Adult Patients with Sickle Cell Disease (SCD)
Acronym: (SCD)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study is terminated prior to its planned completion as anticipated by the protocol due to enrollment completion. Data clean up and analysis is being performed.
Sponsor: Nirmish Shah (Other)
Responsible Party: Sponsor-Investigator, Nirmish Shah, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00110179
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: This will be an open-label, dose escalating study with a starting dose of 2mg. Up to 6 additional cohorts will be enrolled at subsequently higher doses of 4mg, 8mg, 10 mg, 12 mg, 16mg, and 32mg.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AB1 (Experimental): AB1 is the investigational product in this study taken orally, once daily, for 8 weeks. This will be an open-label, dose escalating study with a starting dose of 2mg. Up to 6 additional cohorts will be enrolled at subsequently higher doses of 4mg, 8mg, 10 mg, 12 mg, 16mg, and 32mg.
  Interventions: Drug: AB1

INTERVENTIONS:
Drug: AB1 — This will be an open-label, dose escalating study with a starting dose of 2mg. Up to 6 additional cohorts will be enrolled at subsequently higher doses of 4mg, 8mg, 10 mg, 12 mg, 16mg, and 32mg. Each dose will be taken orally, once daily, for 8 weeks

SUMMARY:
This will be an open-label, dose escalating study with a starting dose of 2mg. Up to 6 additional cohorts will be enrolled at subsequently higher doses of 4mg, 8mg, 10mg, 12mg, 16mg, and 32mg. In each dose escalation cohort, each dose will be taken orally, once daily, for 8 weeks.

DETAILED DESCRIPTION:
This will be an open-label, dose escalating study with a starting dose of 2mg. Up to 4 additional cohorts will be enrolled at subsequently higher doses of 4mg, 8mg, 16mg, and 32mg.

* Cohort 1 - Two (2) patients will be enrolled at the 2mg dose level for 8 weeks of treatment. After both patients have received at least 4 weeks of treatment, if there are no adverse events ≥Grade 2 that are related (possibly, probably, or definitely) to the study drug, then the study will proceed to the next dose level. Note that if ≥Grade 2 toxicity is seen at this dose level, the study drug regimen may be modified (eg, twice or thrice weekly versus daily dosing).
* Cohort 2 - Two (2) patients will be enrolled at the 4mg dose level for 8 weeks of treatment. After both patients have received at least 4 weeks of treatment, if there are no adverse events ≥Grade 2 that are related to the study drug, then the study will proceed to the next dose level.
* Cohort 3 - Three (3) patients will be enrolled at the 8mg dose level for 8 weeks of treatment. After all patients have received at least 4 weeks of treatment, if <2 patients experience a related adverse event ≥Grade 2, then the study will proceed to the next dose level. (If ≥2 patients experience a related adverse event ≥Grade 2, the previous cohort will be expanded.)
* Cohort 4 - Three (3) patients will be enrolled at the 10mg dose level for 8 weeks of treatment. After all patients have received at least 4 weeks of treatment, if <2 patients experience a related adverse event ≥Grade 2, then the study will proceed to the next dose level. (If ≥2 patients experience a related adverse event ≥Grade 2, the previous cohort will be expanded.)
* Cohort 5 - Three (3) patients will be enrolled at the 12mg dose level for 8 weeks of treatment. After all patients have received at least 4 weeks of treatment, if <2 patients experience a related adverse event ≥Grade 2, then the study will proceed to the next dose level. (If ≥2 patients experience a related adverse event ≥Grade 2, the previous cohort will be expanded.)
* Cohort 6 - Three (3) patients will be enrolled at the 16mg dose level for 8 weeks of treatment. After all patients have received at least 4 weeks of treatment, if <2 patients experience a related adverse event ≥Grade 2, then the study will proceed to the next and final dose level. (If ≥2 patients experience a related adverse event ≥Grade 2, the previous cohort will be expanded.)
* Cohort 7 - Three (3) patients will be enrolled at the 32mg dose level for 8 weeks of treatment.
* An additional cohort may be explored at the 24mg dose level if deemed appropriate based on safety and activity parameters.

If there are any adverse events Grade ≥2 that are related (possibly, probably, or definitely) to study drug, at the 4mg cohort or in ≥2 patients in any subsequent cohort, the dose may be reduced to the previous cohort and an additional 3-6 patients (total of up to 9) may be enrolled into that cohort. Additionally, if Hbf levels increase >15% (expressed as a percentage of total Hb) in any cohort, the cohort can be expanded to an additional 3 to 6 patients as well as continue to the next cohort if safety parameters have been met. In the expansion cohort, patients will receive study drug treatment for an additional 4 weeks (total of 12 weeks)..

Approximately 6 to 39 patients may be enrolled for the entire study. Patients are eligible to enroll in a higher cohort of the study after a minimum of one-month washout from AB1 dosing, if their HbF levels return to baseline (<15%) and the investigator deems the patient eligible.

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent
2. Age 18 to 45 years of age, inclusive at screening
3. Confirmed SS or S-b0-thalassemia SCD
4. Sickle crisis rate of 2-10 within the past year with no crisis in the last 28 days
5. HbF <8.6% of total Hb at screening
6. Regular compliance with comprehensive care and previous therapy -

Exclusion Criteria:

1. Experienced severe sepsis or septic shock within the previous 12 weeks
2. Febrile illness in the 1 week prior to baseline visit
3. Acute complications due to SCD (i.e., hospitalization, acute pain, or acute chest syndrome) in the 28 days prior to screening visit
4. Plans for hospitalization, surgery, or other major procedures during the duration of the study or between screening and baseline
5. ALT ≥2X the upper limit of normal or albumin <2.0 mg/dL or direct (conjugated) bilirubin ≥ 1.5 mg/dl*
6. Serum creatinine >2.9 mg/dL and calculated creatinine clearance <30 mL/min# *
7. Platelet count >800 x 109/L OR <150 x 109/L*
8. Absolute neutrophil count <1.5 x 109/L*
9. Currently pregnant or breastfeeding
10. Female of active childbearing potential$ who is unwilling or unable to adhere to the contraception requirements specified in the protocol
11. Male with female partner(s) of childbearing potential$ who is unwilling or unable to adhere to the contraception requirements specified in the protocol
12. Altered mental status or recurrent seizures requiring anti-seizure medications
13. Moribund or any concurrent disease (e.g., hepatic, renal, cardiac, metabolic) of such severity that death within 24 weeks is likely
14. Concurrent diagnosis of malignancy including MDS, leukemia, or an abnormal karyotype
15. Known Vitamin-B12, folate, or iron deficiency
16. New York Heart Association (NYHA) class III/IV status
17. Eastern Co-operative Oncology Group (ECOG) performance status ≥3
18. Participant is on chronic transfusion therapy (e.g., for history of TIA or stroke) and medically contraindicated to discontinue transfusions (unless multiple allo-antibodies prevent the patient from getting transfusions as scheduled)
19. Blood transfusion in the 28 days prior to screening visit or between screening and baseline visits
20. Known history of illicit drug or alcohol abuse within the past 12 months.
21. Current treatment with Oxbryta or Adakveo (must be off therapy for 30 days for Oxbryta with no plans to restart and off therapy for 3 months for Adakveo with no plans to restart)
22. Other experimental or investigational drug therapy in the past 28 days -

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events/serious adverse events as measured by patient report/medical records | From the time of consent up to 12 months
Number of ≥Grade 2 study related adverse events as measured by patient report/medical record | From the time of consent up to 12 months
  Adverse events that cause enough discomfort to interfere with usual daily activity; may warrant therapeutic intervention

SECONDARY OUTCOMES:
Change in Cmax as measured by blood test | Baseline, week4, week8, week10
Change in tmax as measured by blood test | Baseline, week4, week8, week10
Change in t1/2 as measured by blood test | Baseline, week4, week8, week10
Change in AUC o-t as measured by blood test | Baseline, week4, week8, week10
Change in dose normalized AUC o-inf as measured by blood test | Baseline, week4, week8, week10
Change in CL as measured by blood test | Baseline, week4, week8, week10
Change in Vz as measured by blood test | Baseline, week4, week8, week10
Change in Vss as measured by blood test | Baseline, week4, week8, week10
Change in percentage of total percentage of total hemoglobin (HB) as measured by HPLC | Screening, baseline, week2,week4, week6, week8, week10, week12
Change in percentage of F-cells measured by flow cytometry | Screening, baseline, week2,week4, week6, week8, week10, week12
Change in percent reticulocytes as measured by blood tests | Screening, baseline, week2,week4, week6, week8, week10, week12

CONTACTS AND LOCATIONS:
Overall Officials: Nirmish Shah, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Augusta University Medical Center, Augusta, Georgia
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: No